CLINICAL TRIAL: NCT06458686
Title: Effect of Vitamin D Supplementation on Mental Health: An Exploratory Study on A University Students Suffering From Vitamin D Deficiency
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: German University in Cairo (Other)
Collaborators: Prof. Mohamed Hassan Solayman, Clinical pharmacy Department, German University in Cairo (Unknown); Prof. May Ahmed Shawki, Clinical Pharmacy Department, Ain Shams University, Egypt (Unknown)
Responsible Party: Principal Investigator, Nouran Hussien Kandeel, Nouran hussien kandeel, German University in Cairo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1234
Record Dates: First submitted 2024-06-09; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Psychiatric Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): This group does not take any drug. It will take placebo.
  Interventions: Other: Placebo
- Intervention group (Active Comparator): This group will take Vitamin D
  Interventions: Drug: Vit D

INTERVENTIONS:
Drug: Vit D — Vitamin D is a fat soluble vitamin used for the treatment of many diseases.
  Arms: Intervention group
Other: Placebo — Placebo is a non drug formulation
  Arms: Control group

SUMMARY:
University students are susceptible to psychological burdens such as depressive symptoms, anxiety, and stress which might have been linked to vitamin D deficiency. Low serum vitamin D level is well recognized around the world. Vitamin D has been reported to modulate several neurological pathways in the brain that control psychological function. As a result, the purpose of this study is to evaluate the effect of vitamin D supplementation on the presence of depressive symptoms, anxiety, and stress in university students. The study will include two phases. The first phase is a cross-sectional phase assessing the prevalence vitamin D deficiency in addition to psychological symptoms. The second phase is a randomized controlled clinical trial that aims to assess the effect of vitamin D supplementation on the prevalent psychological symptoms and its impact on the academic performance among university students. The study will look at the relationship between mental health and vitamin D deficiency, as well as how it will affect academic performance of university students.

ELIGIBILITY:
Inclusion Criteria:

* For phase 1: sample will be selected using convenient sampling method where all students with an age range 18-22 years old fulfilling the eligibility criteria will be educated about the study protocol and will be asked to participate in the study.

For phase 2: students who diagnosed with deficient vitamin D level will be asked to participate in the study.

Exclusion Criteria:

* Hypersensitivity to oral vitamin D supplements such as Diviton or Vidrop.

  * Students taking medications affecting vitamin D metabolism such as anti-seizure medications: phenytoin, phenobarbital and carbamazepine, isotretinoin, steroids: dexamethasone, antibiotics: isoniazid and rifampin and antifungals: clotrimazole.
  * Students taking antidepressants, drug for bipolar disorder treatment like lithium and antipsychotic agents like olanzapine.
  * Students with insufficient vitamin D level (20-30 ng/mL).
  * Students with confirmed diagnosis with psychiatric illness.
  * Students with a history of liver disease or dysfunction.
  * Students with a history of kidney disease or dysfunction.

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the correlation between vitamin D deficiency and presence and severity of anxiety, stress and depressive symptoms. | 3 months
  Evaluation of the correlation between vitamin D deficiency and presence and severity of anxiety, stress and depressive symptoms.